CLINICAL TRIAL: NCT06592170
Title: A Single Arm, Open Center, Multicenter Clinical Study of Frontline Treatment of Marginal Zone Lymphoma Patients (MZL) With Linperlisib Combined With Obinutuzumab
Brief Title: Linperlisib Combination With Obinutuzumab Frontline Treatment of Marginal Zone Lymphoma Patients (MZL)
Acronym: MZL-001
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Ou Bai, MD/PHD, Director, The First Hospital of Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YY-20394-MZL-001
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Safe import period: Linperlisib: 80 mg, oral (pre - and post meal), QD; obinutuzumab: 1000 mg, intravenous infusion, administered on the first day (1st cycle on days 1, 8, and 15); Every 28 days, there is one cycle in total.
  Extended treatment period: Combination induction: Linperlisib: RP2D, oral (pre - and post meal), QD; obinutuzumab: 1000 mg/time, intravenous infusion, administered on the first day (1st cycle on days 1, 8, and 15); Every 28 days, there are 2 cycles in total. Afterwards, single drug maintenance: Linperlisib: RP2D, oral (before and after meals), QD; every 28 days per cycle.
  Interventions: Drug: Linperlisib combination with obinutuzumab

INTERVENTIONS:
Drug: Linperlisib combination with obinutuzumab — Safe import period: Linperlisib: 80 mg, oral (pre - and post meal), QD; obinutuzumab: 1000 mg, intravenous infusion, administered on the first day (1st cycle on days 1, 8, and 15); Every 28 days, there is one cycle in total.
  Extended treatment period: Combination induction: Linperlisib: RP2D, oral (pre - and post meal), QD; obinutuzumab: 1000 mg/time, intravenous infusion, administered on the first day (1st cycle on days 1, 8, and 15); Every 28 days, there are 2 cycles in total. Afterwards, single drug maintenance: Linperlisib: RP2D, oral (before and after meals), QD; every 28 days per cycle.

SUMMARY:
This is a single arm, open label, national multicenter clinical study included patients with marginal zone lymphoma patients (MZL) , aim is to evaluate the efficacy and safety of first-line treatment with Linperlisib combined with obinutuzumab in patients with marginal zone lymphoma (MZL).

DETAILED DESCRIPTION:
This study is a single arm, open label, multicenter Phase Ib/II study aimed at evaluating the safety and efficacy of first-line treatment of patients with marginal zone lymphoma with combination therapy of Linperlisib and obinutuzumab. The study is divided into Phase Ib safety introduction stage, and Phase II is recommended; As well as the Phase II expansion phase, the research design is shown in the following figure. Phase Ib is the safety introduction period, with the main purpose of determining the recommended Phase II effective dose (RP2D) based on dose limiting toxicity (DLT). Six subjects are planned to be enrolled to observe the safety of one cycle of combination therapy with Linperlisib (80 mg, once daily). If<2 cases of DLT occur, the RP2D of Linperlisib will be 80 mg, once daily; If there are ≥ 2 cases of DLT, RP2D is 60 mg once daily. Phase II is the expansion phase, which involves induction therapy with two cycles of Linperlisib RP2D combined with obinutuzumab. All patients who achieve complete remission (CR) or partial remission (PR) after induction therapy receive induction therapy with a dose of Linperlisib, which is maintained every 28 days for one cycle until disease progression or other reasons lead to discontinuation. During the maintenance phase, the use of Linperlisib should not exceed 24 months. If the disease is stable (SD) or (PD), the patient will be removed from the group. If a patient fails to achieve CP or PR after two cycles of induction therapy, the researcher will determine whether to continue induction therapy. Induction therapy can last up to six cycles.The aim is to evaluate the efficacy and safety of first-line treatment with Linperlisib combined with obinutuzumab in patients with marginal zone lymphoma (MZL).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years old, both male and female are acceptable; 2. Newly diagnosed marginal zone lymphoma confirmed by histopathology. Including extranodal MZL, intranodal MZL, and splenic MZL; 3. There is at least one measurable lesion: the longest diameter (LDi) of a lymph node lesion is greater than 1.5 cm or the LDi of an extra lymph node lesion is greater than 1 cm (according to the 2014 Lugano classification); 4. The physical status score of the Eastern Cooperative Oncology Group (ECOG) is ≤ 2; 5. Expected lifespan ≥ 12 weeks; 6. Have not received any previous anti-tumor treatment; 7. Possess sufficient bone marrow and organ functions; 8. All screening laboratory tests must be conducted according to the protocol requirements, and must be conducted within 7 days prior to enrollment. The values of laboratory tests conducted for screening must meet the following standards:

Blood routine examination (no blood transfusion within 14 days before screening, no use of granulocyte colony-stimulating factor (G-CSF), no medication correction):

1. Hemoglobin (Hb) ≥ 90 g/L;
2. Neutrophil count (ANC) ≥ 1.5 × 10*9/L;
3. Platelets (PLT) ≥ 100 × 10*9/L;

Biochemical examination:

1. TBIL<1.5 x upper limit of normal range (ULN);
2. Glutamate alanine aminotransferase (ALT) and Glutamate aspartate aminotransferase (AST) ≤ 2.5 × ULN;
3. Serum creatinine (Cr) ≤ 1.25 × ULN or Endogenous creatinine clearance rate ≥ 60 mL/min (Cockcroft Gault formula);

Coagulation function:

1. International Normalized Ratio (INR) ≤ 1.5 × ULN;
2. Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; 9. Women who have the possibility of pregnancy must undergo a serum pregnancy test within 7 days before the first use of the test drug, and the result must be negative. They must also be willing to use effective contraception methods during the trial period and within 1 year after the last administration of the test drug. For male participants whose partners are women of childbearing age, surgical sterilization should be performed, or they should agree to use efficient contraception methods during the trial period and one year after the last administration of the trial drug; 10. The subjects voluntarily joined this study, signed an informed consent form, had good compliance, and cooperated with follow-up

Exclusion Criteria:

* 1. Patients who have received any targeted PI3K therapy before enrollment; 2. History of other primary invasive malignant tumors that have not been relieved or have not been relieved for more than 3 years; 3. Patients with involvement of the central nervous system (meninges or brain parenchyma); 4. Individuals who are known to have allergies to any of the drugs in the study; 5. Participated in clinical trials of other drugs within 4 weeks prior to the start of the study; 6. Pregnant or lactating women; 7. Individuals with active infections, except for those with tumor related B symptoms and fever; 8. Combined diseases and medical history:

  1. There are multiple factors that can affect oral medication, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
  2. Individuals with a history of abuse of psychotropic drugs who are unable to quit or have mental disorders;
  3. Subjects with any severe and/or uncontrolled illnesses, including:

     1. Poor blood pressure control (systolic blood pressure ≥ 150mmHg or diastolic blood pressure ≥ 100 mmHg);
     2. Suffering from ≥ grade 2 myocardial ischemia or myocardial infarction, arrhythmia [including QTc ≥ 450ms (male), QTc ≥ 470ms (female)], and ≥ grade 2 congestive heart failure [New York Heart Association (NYHA) classification];
     3. Active interstitial pneumonia or other chronic lung diseases leading to severe impairment of lung function, defined as FEV1 and DLCOc<60% of normal predicted values; History of interstitial pneumonia caused by COVID-19.
     4. Liver abnormalities:
     5. Decompensated cirrhosis (Child Pugh liver function rating B or C)
     6. Known history of liver disease with clinical significance. Including viral hepatitis, known carriers of hepatitis B virus (HBV) must exclude active HBV infection, i.e. HBV DNA positive (>2500 copies/mL or >500IU/mL, and greater than the upper limit of normal); Known to be infected with hepatitis C virus (HCV) and HCV RNA positive (>1 × 103 copies/mL). Note: hepatitis B HBsAg positive subjects who meet the inclusion conditions, whether their HBV DNA is measurable or not, need to continue antiviral treatment (nucleoside analogues are recommended) and regularly monitor HBV DNA; For subjects with positive HBcAb but negative HBsAg in hepatitis B, HBV DNA should be monitored regularly and preventive antiviral treatment should be recommended; HCV RNA should be regularly monitored in subjects with hepatitis C.
     7. Patients with renal failure requiring hemodialysis or peritoneal dialysis;
     8. Subjects with uncontrolled pleural effusion, pericardial effusion, or ascites that require repeated drainage;
     9. Poor control of diabetes (FBG>10mmol/L);
     10. Urine routine shows urinary protein ≥++and confirms 24-hour urinary protein quantification>1.0g; 9. History of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation; 10.According to the researchers assessment, there are accompanying diseases that pose a serious threat to patient safety or affect the completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-08-13 (Estimated); Study Completion 2027-08-13 (Estimated)

PRIMARY OUTCOMES:
Complete response（CR） according to the RECIST 1.1 | 6 months from the start of linperlisib treatment
  The CR rate of patients with Linperlisib in combination with Obinutuzumab for marginal zone lymphoma

SECONDARY OUTCOMES:
Objective Response Rate (ORR) according to the RECIST 1.1 | 6 months from the start of linperlisib treatment
  The ORR rate of patients with Linperlisib in combination with Obinutuzumab for marginal zone lymphoma
Duration of Overall Response (DOR） | Within 2 year from the start of Linperlisib treatment，the time from the first judgment of complete remission (CR) or partial remission (PR) to the discovery of disease progression (PD)
  The time from the first judgment of complete remission (CR) or partial remission (PR) to the discovery of disease progression (PD).
Adverse event | Within 2 year from the start of Linperlisib treatment
  Refers to adverse medical events that occur in the clinical trial process of the subject
Disease control rate（DCR） | Within 2 year from the start of Linperlisib treatment
  Proportion of patients with remission (PR+CR) and stable disease (SD) within 2 years after Linperlisib treatment.
Progression-free survival（PFS） | Within 2 years of initiation of Linperlisib treatment
  The time from the start of clinical trials to the occurrence (in any aspect) of tumor progression or death due to any reason

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No